CLINICAL TRIAL: NCT05006027
Title: Feasibility of Percutaneous Coronary Intervention Using a 7-Fr Thin Walled Sheath Via the Distal Radial Approach: a Prospective Observational Study (SEVEN-BOX)
Brief Title: Feasibility of PCI Using a 7-Fr Thin-Walled Sheath Via the DRA
Acronym: SEVEN-BOX
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Collaborators: Severance Hospital (Other); Merit Medical Systems, Inc. (Industry)
Responsible Party: Principal Investigator, Yongcheol Kim, Director head of snuffbox center in Yongin Severance Hospital, Principal Investigator, Clinical Professor, Yonsei University
Other Study IDs: 9-2021-0031
Record Dates: First submitted 2021-08-08; First posted 2021-08-16 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease; Distal Radial Artery; Complex Intervention
Keywords: distal radial artery; coronary artery disease; percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Percutaneous coronary intervention using a 7-Fr thin-walled sheath via the distal radial approach: patients with coronary artery disease who planned to perform PCI using 7-Fr thin-walled sheath via the distal radial approach
  Interventions: Procedure: Percutaneous coronary intervention via the distal radial approach

INTERVENTIONS:
Procedure: Percutaneous coronary intervention via the distal radial approach — Percutaneous coronary intervention using a 7-Fr thin walled sheath (Prelude IDeal, MERIT MEDICAL, South Jordan, UT, USA) via the distal radial approach

SUMMARY:
To evaluate the safety and effectiveness of percutaneous coronary intervention using a 7-French(Fr) thin-walled sheath via the distal radial approach

DETAILED DESCRIPTION:
Recently, coronary angiography (CAG) and percutaneous coronary intervention (PCI) via the distal radial artery access (DRA) have shown several advantages owing to fewer complications, such as radial artery occlusion, pseudoaneurysms, and arteriovenous(AV) fistulas, and short hemostasis duration than the proximal radial access (PRA). However, despite the potential advantages of the DRA, there are still many cardiologists who prefer the femoral approach for complex PCI including left main disease, bifurcation lesions, heavily calcified lesions, which need a strong backup and using several devices. The radial artery and the distal radial artery have a smaller diameter than the femoral artery, and interventional cardiologists are usually performed using the 6-Fr sheath. The previously developed 7-Fr sheath has a higher risk of vascular occlusion when use in a radial artery due to larger diameter compared to radial artery in 30% to 60% of patients. However, with the recent development of various technologies, the outer diameter of the sheath is gradually becoming thinner and recently a 7-Fr thin-walled sheath which does not differ significantly from the outer diameter of the 6-Fr sheath used in the previously PRA demonstrated that feasibility and safety for radial artery intervention. Despite the feasibility and potential benefits of the DRA and 7-Fr thin-walled sheath for radial artery, there is a lack of data regarding the safety and efficacy of a 7-Fr thin-walled sheath during the DRA.

ELIGIBILITY:
Inclusion Criteria:

* Patients, ≥ 19 years of age, who were diagnosed with ischemic heart disease requiring percutaneous coronary intervention (PCI)
* Patients who are palpable distal radial artery
* The decision to participate voluntarily in this study and the written consent of the patient
* Patients who planned to perform PCI using a 7-Fr thin-walled sheath

Exclusion Criteria:

* Patients who are not palpable distal radial artery
* Female of childbearing potential, who possibly plans to become pregnant any time after enrollment into this study
* Pregnancy
* Patients who are not appropriate for this study

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with coronary artery disease who planned to perform PCI using a 7-Fr thin-walled sheath will be recruited
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Access site complication during hospitalization and within 1-month follow-up | Through procedure completion, up to 1month
  bleeding(defined by BARC criteria), hematoma (using modified EASY[Early Discharge After Transradial Stenting of Coronary Arteries Study] classification: A) Grade Ia hematoma was subclassiﬁed into 4 grades from the puncture site [Grade 1, <2cm; Grade2, 2-5cm; Grade3,>5cm; and grade 4, hand swelling], B) Grade Ib, wrist < 5cm, C) Grade II, wrist < 10cm, D) Grade III, forearm, E) Grade IV, upper arm), numbness, AV fistula, Pseudoaneurysm, and conventional and distal radial artery occlusion (assessed by manual palpation or ultrasonography[prefer])
Success rate of PCI | Through procedure completion, up to 1month
  Success rate of PCI using 7-Fr sheath via the distal radial approach (%)

SECONDARY OUTCOMES:
Hemostasis duration | Through procedure completion, up to 24 hours
  Hemostasis duration using 7-Fr thin-walled sheath via the distal radial approach (minute)
Patency of proximal radial artery after hemostasis | Through procedure completion, up to 24 hours
  Patency of proximal radial artery using 7-Fr thin-walled sheath via the distal radial approach by ultrasonography after hemostasis (%)
Patency of distal radial artery after 1 month | Time Frame: up to 1month
  Patency of distal radial artery using 7-Fr thin-walled sheath via the snuffbox approach by ultrasonography after 1-month (%)

OTHER OUTCOMES:
If intravascular imaging modalities (OCT/IVUS) are seen during intervention, check for conventional radial radial artery complications through OCT/IVUS | Through procedure completion
  If intravascular imaging modalities (OCT/IVUS) are seen during intervention, check for conventional radial radial artery complications through OCT/IVUS

CONTACTS AND LOCATIONS:
Overall Officials: Yongcheol Kim, MD, Principal Investigator — Yongin Severance Hopistal
Locations (2):
- South Korea (2):
  - Yongin Severance Hospital, Yongin, Gyeonggi-do
  - Yongin Severance Hospital, Yŏngin

IPD SHARING:
Plan to Share IPD: No
No planned

REFERENCES:
- [Derived] Roh JW, Lee OH, Heo SJ, Kim Y, Im E, Cho DK. Feasibility of percutaneous coronary intervention using a 7-French thin-walled sheath via the distal radial access. Sci Rep. 2025 May 15;15(1):16961. doi: 10.1038/s41598-025-01149-1. PMID 40374669